CLINICAL TRIAL: NCT02474212
Title: Anti-Xa Concentrations With Continuous Intravenous Infusion and Subcutaneous Administration of Enoxaparin After Coronary Artery Bypass Grafting: Randomized Clinical Trial
Brief Title: : Pharmacokinetics of Enoxaparin After Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Heart Hospital, Tampere University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 290115-1
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism; Thromboprophylaxis
Keywords: Venous thromboembolism; pulmonary embolism; thromboprophylaxis; anticoagulant; anti-FXa; low-molecular weight heparin; enoxaparin
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Enoxaparin 40 mg s.c. (Active Comparator): Subcutaneous enoxaparin (Klexane®, Sanofi-Aventis) 40 mg thromboprophylaxis every 24 hours for three days (72 hours)
  Interventions: Drug: Enoxaparin
- Enoxaparin 40 mg i.v. (Active Comparator): Enoxaparin thromboprophylaxis (40 mg) daily as continuous intravenous infusion for three days (72 hours)
  Interventions: Drug: Enoxaparin
- Enoxaparin 0.5 mg/kg s.c. (Active Comparator): Subcutaneous enoxaparin (Klexane®, Sanofi-Aventis) 0.5 mg/kg thromboprophylaxis twice a day for three days (72 hours)
  Interventions: Drug: Enoxaparin
- Enoxaparin 1 mg/kg i.v. (Active Comparator): Enoxaparin thromboprophylaxis 1 mg/kg daily as continuous intravenous infusion for three days (72 hours)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
To evaluate the pharmacokinetics of thromboprophylactic doses of LMWH enoxaparin in postoperative CABG patients, drug is administered either as a continuous intravenous infusion (CIV) or subcutaneous bolus (SCB) once per 72h. Plasma anti-Xa values are measured 12-14 times during study period and concentration maximums calculated to enable comparison of anti-Xa values between administration routes.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled trial. After informed consent, 80 elective on pump CABG patients with a clinical indication for post-operative thromboprophylaxis will be studied in the Tampere University Heart Hospital. Study has two independent parts with 40 patients in both. Results are reported separately from these two parts of the study.

Firts part of the study: After written consent, 20+20 patients are randomized to receive enoxaparin either as continuous intravenous infusion (treatment group) or subcutaneous bolus injection (control group). Enoxaparin dose is 40mg/24h either CIV of SCB. Anti-Xa values are measured 12-14 times from blood samples to evaluate the anticoagulation effect of enoxaparin.

Second part of the study: After written consent, 20+20 patients are randomized to receive enoxaparin either as continuous intravenous infusion (treatment group) or subcutaneous bolus injection (control group). Enoxaparin dose is 1mg/kg/24h in CIV group and 0,5mg/kg twice a day in SCB group. In this second part of the study with eleveted enoxaparin dosage, 4 additional blood samples will be taken and analysed by ROTEM to investigate the overall coagulation status of the patients before and after the initiation of enoxaparin.

The study will consist of two independent parts.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-33 kg/m2
* Elective on-pump CABG operation
* Indication for post-operative pharmacological thromboprophylaxis
* Written informed consent obtained from the patient or his/her legal representative.

Exclusion Criteria:

* Other indications for anticoagulant therapy than thromboprophylaxis
* Known heparin induced thrombocytopenia (HIT), or hypersensitivity to enoxaparin or heparin
* Any long-term anticoagulant medication, expect low-dose aspirin
* Major bleeding within the last week unless definitively treated
* Blood platelet count <20, P-TT <20 % or INR >1.7
* GFR less than 30 ml/min/1.73 m2 estimated from serum creatinine by applying Cockcroft-Gault equation 13 or chronic dialysis
* Known HIV, HBV, or HCV infection
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Anti-Xa concentration maximum 0-24h (Cmax0-24h) | 0-24h after initiation of enoxaparin
  Anti-Xa concentration maximum level calculated from measured values during 0-24h after initiation of enoxaparin.

SECONDARY OUTCOMES:
Anti-Xa concentration maximum 25-72 h (Cmax25-72h) | 25-72 h after initiation of enoxaparin
  Anti-Xa concentration maximum level calculated from measured values 25-72h after the initiation of enoxaparin.
Anti-Xa trough concentartion at 72 h (C72h) | 72 h after the initiation of enoxaparin
  Anti-Xa concentration at the of 72h study period

OTHER OUTCOMES:
Clinical outcomes | 0-90 days after initiation of enoxaparin
  Postoperative bleeding, DVT, pulmonary embolism, 90 day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland